CLINICAL TRIAL: NCT03220607
Title: The Predictive Performance of Uterocervical Angle in the Termination of Second Trimester Pregnancy
Brief Title: Uterocervical Angle in the Termination of Second Trimester Pregnancy
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Berna Aslan Cetin, MD,ObGYN, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2016/5
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Abortion, Second Trimester
Keywords: uterocervical angle, second trimester abortion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Medical induced abortion: 120 singleton nulliparous patients are planning to complete the study period. Study group constitute of second trimester pregnancies between 14-24 weeks of gestation. All participants were nulliparous and had no systemic illnesses. The uterocervical angle will be measured in all participants before the induction of labor.
  Interventions: Other: uterocervical angle

INTERVENTIONS:
Other: uterocervical angle — uterocervical angle is the angle between lower segment of uterus and cervix

SUMMARY:
To evaluate the performance of uterocervical angle (UCA) in the prediction of second trimester terminations.

DETAILED DESCRIPTION:
Medical termination of pregnancy is a common procedure in obstetrics. In recent years, uterocervical angle (UCA) emerged as a new ultrasound parameter in the prediction of labor. Dziadosz et al concluded that the performance of UCA was even better than the cervical length in their cohort. A wide UCA during second trimester shown to have an increased risk of preterm labor and narrow angle was less likely to have labor.

The investigators are aimed to investigate predictive role of both cervical length and UCA in the termination of second trimester pregnancy.The investigators focused on nulliparous women who are taking misoprostol for the cervical preparation and aim to measure their UCA.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous singleton pregnancy
* no previous systemic illnesses

Exclusion Criteria:

* abnormal Pap smear
* previous cesarean section
* history of dilatation and curettage (D&C)
* history of LEEP and cervical conization

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant population undergoing second trimester abortion
Study Population: Pregnant population undergoing medical induced second trimester abortion.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2016-10-15 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
uterocervical angle | once at the beginning of enrollment
  the angle between the lower segment of uterus and cervix

CONTACTS AND LOCATIONS:
Overall Officials: Alev Atis, MD,ObGyn, Study Director — Kanuni Sultan Suleyman Training and Research Hospital
Locations (1):
- Kanuni SSTRH, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Uterocervical angle: a novel ultrasound screening tool to predict spontaneous preterm birth. — http://www.ncbi.nlm.nih.gov/pubmed/27018466